CLINICAL TRIAL: NCT02190643
Title: Improving Nicotine Patch Adherence Among Latino HIV-Positive Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21DA035629 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Smoking
Keywords: Smoking; HIV; Latino; Cessation; Nicotine patch
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adherence condition (Experimental): Brief smoking cessation counseling session (based on 5 A's approach) that includes a module focused on improving adherence to using the nicotine patch, plus 8-week supply of nicotine patches.
  Interventions: Behavioral: Cessation counseling with adherence focus
- Standard condition (Active Comparator): Brief smoking cessation counseling session (based on 5 A's approach) that does not include a module focused on improving nicotine patch adherence, plus 8-week supply of nicotine patches.
  Interventions: Behavioral: Cessation counseling without adherence focus

INTERVENTIONS:
Behavioral: Cessation counseling with adherence focus
  Arms: Adherence condition
Behavioral: Cessation counseling without adherence focus
  Arms: Standard condition

SUMMARY:
The goal of this study is to evaluate a smoking cessation program for Latino HIV-positive smokers focused on improving adherence to using the nicotine skin patch.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Latino
* HIV positive
* current, daily smoker
* ready to set quit date in next 30 days
* willing to try the nicotine patch

Exclusion Criteria:

* suffering from any medical condition which would prevent using the nicotine patch
* currently using other tobacco products or e-cigarettes
* currently receiving counseling or medication to quit or reduce smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence | 3 months post-quit date
  No smoking from the target quit date through the 3-month follow-up
biochemically-verified 7-day point prevalence abstinence | 3 months post-quit date
  No smoking in the 7 prior days

SECONDARY OUTCOMES:
Nicotine patch adherence | 3 months post-quit date

CONTACTS AND LOCATIONS:
Locations (1):
- Bienestar Human Services Inc, Los Angeles, California, United States